CLINICAL TRIAL: NCT07248488
Title: Effect of an Intervention Combining the Use of Standardized Information and Sending an SMS Advice Message to Parents Calling the SAMU Center 15 for Uncomplicated Fever in Children Over 3 Months and Under 10 Years of Age : a Regional Cluster Randomized Trial
Brief Title: Effect of an Intervention Combining the Use of Standardized Information and Sending an SMS Advice Message to Parents Calling the SAMU Center 15 for Uncomplicated Fever in Children
Acronym: SCF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-07
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Emergency Call; Fever; Pediatric Fever Management; Parental Anxiety
MeSH Terms: conditions — Fever

STUDY DESIGN:
Intervention Model Description: Randomized controlled cluster trial, open-label, in the AuRA region, evaluating the superiority of using a standardized protocol for regulating fever in children, combining systematic recommendations and sending an SMS with advice to parents, compared to current practice (no standardized protocol, no text message advice) on the rate of unscheduled healthcare visits 7 days after the initial call to the 15 emergency center.
  In both arms of the study, unscheduled healthcare visits within 7 days of the initial call will be assessed by responses to the follow-up text message on day 7 and a phone call from a Center 15 doctor between days 14 and 21, if the child has been hospitalized.
  All patients included in the study will be followed up for a minimum of 7 days and a maximum of 21 days after the initial call to the 15 Center.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combined intervention (Experimental): Standardized recommendations during emergency calls and sending of advisory text messages
  Interventions: Other: Standardized recommendations during emergency calls and sending advisory text message
- Traditional regulation (No Intervention)

INTERVENTIONS:
Other: Standardized recommendations during emergency calls and sending advisory text message — When the emergency service is called, the coordinating physician provides standardized recommendations based on the treatment guidelines issued by the French Pediatric Society. After the emergency call, the parent who made the call receives a text message summarizing all the advice given by the doctor.
  Arms: Combined intervention

SUMMARY:
During the winter of 2022/23, a standardized protocol for managing fever in children aged 3 months to 10 years was implemented at Annecy Genevois Hospital for a period of one month. This protocol included advice given by the regulator and sending a text message to parents after the call. A total of 182 calls were handled in one month: 95 during a 15-day period before the intervention was rolled out and 87 during a 15-day period during the intervention (43 with unread text messages and 44 with read text messages). All parents who read the text message understood it. The rate of compliance with advice was improved by the intervention when the text message was read (p < 0.01), in terms of increased paracetamol intake, avoidance of cold baths, undressing the child, and administering fluids. When the text message was read, the rate of calls to the 15 emergency center fell from 13% before the intervention to 2% when the text message was read (p = 0.04). A downward trend in emergency room visits was also observed, from 13% before the intervention to 5% when the text message was read and 19% when the text message was not read (p = 0.13). These encouraging data suggest that a randomized study would demonstrate the value of this approach in routine practice.

Even if the effect of such protocols is moderate, the target audience is such that their impact on the use of unscheduled care and on the healthcare system could be significant, at a low implementation cost.

The use of a standardized protocol involving the sending of text messages in cases of uncomplicated fever in children makes it possible to:

* standardize the advice given by call center doctors,
* ensure the traceability of advice,
* help parents monitor their children.

The objective of this study is to determine, in a randomized trial, whether the combined use of standardized advice for children with fever and text messages sent to parents by the emergency medical service (EMS) can:

i) reduce the use of unscheduled medical care; ii) improve compliance with advice; iii) reduce the rate of callbacks to the emergency medical service; iv) improve parent satisfaction.

ELIGIBILITY:
Inclusion criteria relating to the child concerned by the call to the SAMU Centre 15:

* Call for a child aged between 3 months and 10 years,
* Presenting with fever alone (SFMU/GPIP definition),
* Developing for less than 72 hours,
* Without clinical signs,
* And without signs of seriousness requiring emergency medical attention (as determined by SAMU Centre 15):

  * Fever ≥41°C,
  * Impaired consciousness,
  * Convulsions,
  * Dyspnea,
  * Skin rash,
  * Dehydration.

Inclusion criteria relating to the caller:

* Caller with parental authority over the child concerned by the call,
* Affiliated to a social security scheme or beneficiary of a similar scheme.

Exclusion criteria relating to children involved in calls to the SAMU Centre 15 emergency medical service:

* Children who have already been the subject of a call to the SAMU Centre 15 emergency medical service in the last 15 days,
* Children with a history of urinary tract infection,
* Children referred by the dispatcher during the phone call to a healthcare facility for clinical evaluation (SMUR, private ambulance, fire department, parents referred to the emergency room or primary care physician).

Exclusion criteria relating to the caller:

* Calls made from a landline or foreign number, making it impossible to send text messages,
* Calls made by someone who cannot read or understand French.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1792 (Estimated)
Dates: Start 2026-09-07 (Estimated); Primary Completion 2028-03-20 (Estimated); Study Completion 2028-03-28 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of a standardized protocol for managing childhood fever, combining systematic recommendations and text messages sent to parents with advices on seeking unscheduled care: visits to the emergency room and/or medical consultations | 21 days after the initial emergency call to the SAMU Centre 15

CONTACTS AND LOCATIONS:
Overall Officials: Virginie SAVRY, MD, Principal Investigator — Centre Hospitalier Annecy Genevois
Locations (1):
- CH Annecy Genevois, Annecy, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No